CLINICAL TRIAL: NCT03119688
Title: A Clinical Study to Assess the Mildness of a Cosmetic Cleanser in Healthy Subjects Using the Forearm-Controlled Application Technique (FCAT)
Brief Title: To Assess the Mildness of a Cosmetic Cleanser in Healthy Participants Using the Forearm-Controlled Application Technique (FCAT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 207619
Record Dates: First submitted 2017-04-05; First posted 2017-04-18 (Actual); Results first posted 2019-05-02 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-01

CONDITIONS: Skin Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Test product (Other): 0.09 milliliters (ml) of the cleanser (test product) will be applied on the allocated site on forearm topically.
  Interventions: Other: Test Product
- Positive Control (Other): Soap bar (positive control) will be applied on the allocated site on forearm by topical dermal administration of towel moistened with sterile water that had been rubbed onto the 100 g bar of soap for 6 seconds to generate a lather.
  Interventions: Other: Positive Control
- Negative Control (Other): 0.09 ml of sterile water (Reference Product) will be applied on the allocated site on forearm topically.
  Interventions: Other: Reference Product
- No Treatment (Other): An area of the forearm that remained unwashed and was included in the study as a reference for the treated areas.
  Interventions: Other: No Treatment

INTERVENTIONS:
Other: Test Product — Micellar cleanser (0.09 ml)
  Arms: Test product
Other: Positive Control — Bar Soap (rubbed for 6 seconds to generate a lather)
  Arms: Positive Control
Other: Reference Product — Sterile Water (0.09 ml)
  Arms: Negative Control
Other: No Treatment — Unwashed area of the forearm
  Arms: No Treatment

SUMMARY:
The objective of this clinical study is to assess the relative mildness of a cosmetic facial cleanser in comparison to water through repeated application to the volar forearm using the FCAT wash procedure.

DETAILED DESCRIPTION:
This is a test site randomized, examiner blinded, positive and negative-controlled, single-center; Forearm Controlled Application Technique clinical study in healthy participants to assess the mildness potential of a cosmetic facial cleansing product.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
* Aged between 18 and 65 years inclusive.
* Good general and mental health with, in the opinion of the investigator or medically qualified designee no clinically significant and relevant abnormalities in medical history or upon physical examination.
* Intact skin at the proposed application site; volar forearm.
* Clinical assessment for eligibility by a dermatologist to ensure participant is free of clinically relevant dermatological conditions.
* Fitzpatrick phototype I to IV.
* Trained examiner scores of zero for dryness and redness for each volar forearm at Screening visit (Visit 1) and each allocated test site on each forearm at Baseline visit.
* Agreement to comply with the procedures and requirements of the study and to attend the scheduled assessment visits.

Exclusion Criteria:

* Women who are known to be pregnant or who are intending to become pregnant over the duration of the study.
* Women who are breast-feeding
* Any history of significant dermatological diseases or conditions or medical conditions known to alter skin appearance or physiologic response (e.g. diabetes,) which could, in the opinion of the Investigator, preclude topical application of the investigational products and/or interfere with the evaluation of the test site reaction.
* Presence of open sores, pimples, or cysts at the application site.
* Active dermatosis (local or disseminated) that might interfere with the results of the study.
* Considered immune compromised.
* History of diseases aggravated or triggered by ultraviolet radiation.
* History of atopic dermatitis.
* Participants with dermatographism.
* Currently using any medication which in the opinion of the investigator, may affect the evaluation of the study product, or place the participant at undue risk.
* Use of the following topical or systemic medications: immunosuppressants, antihistamines, non-hormonal anti-inflammatory drugs, and corticosteroids upto 2 weeks before screening visit.
* Oral or topical treatment with vitamin A acid and/or its derivatives up to 1 month before the screening visit.
* Intention of being vaccinated during the study period or has been vaccinated within 3 weeks of the screening visit.
* Currently receiving allergy injections, or received an allergy injection within 7 days prior to Visit 1, or expects to begin injections during study participation.
* Previous history of atopy, allergic reactions, irritation or intense discomfort feelings to topical-use products, cosmetics or medication.
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Participation in another clinical study (including cosmetic studies) or receipt of an investigational drug within 30 days of the screening visit.
* Previous participation in this study.
* Recent history (within the last 5 years) of alcohol or other substance abuse.
* Intense sunlight exposure or sun tanning sessions, including use of self-tanning products on the test areas up to 14 days before the Screening evaluation.
* Intention of bathing (in the sea or pool), sauna, water sports, or activities that lead to intense sweating.
* Any Participant who, in the judgment of the Investigator and Dermatologist, should not participate in the study.
* Any skin marks on the test site that might interfere with the evaluation of possible skin reactions (e.g. pigmentation disorders, vascular malformations, scars, tattoos, excessive hair, numerous freckles).
* Prisoner or involuntary incarcerated participant
* Participant from an indigenous tribe.
* An employee of the sponsor or the study site or members of their immediate family.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2017-05-26 (Actual); Study Completion 2017-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline; GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- GSK Investigational Site, Campinas, São Paulo, Brazil

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from one center in Brazil.
Pre-assignment Details: A total of 89 participants were screened, out of which 39 participants did not meet the study criteria. Remaining 50 participants were enrolled in the study, out of which 2 participants were not randomized to the study due to adverse events (AEs).
Groups:
- Overall Participants: All participants enrolled in the study received all the study products and received at least 1 wash procedure. Each participant received 9 controlled wash applications over 5 days of test product (0.09 mL), positive control (soap bar) and negative control (0.09 mL) at each allocated test site. Therefore, each participant received a total of 27 applications of study products. Each wash procedure included a 10-second application of the test product, followed by a 90-second wait and a 15-second rinse-off with sterile water.
Period: Overall Study
Arm/Group | Overall Participants
Started | 48
Completed | 44
Not Completed | 4
Not completed — Adverse Event | 4

BASELINE CHARACTERISTICS:
Population: Baseline parameters were reported for safety population. The safety population (N=48) included all participants who had received at least one wash procedure.
Arm/Group | Overall Participants
Number analyzed (Participants) | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.1 (13.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 39
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Visual Assessment of Dryness at Day 5
Description: Skin dryness was assessed by a trained examiner according to following the scoring scale: 0 (No dryness); 1 (Patches of slight powederiness and occasional patches of small scales may be seen, distribution generalized.); 2 (Generalised slight powederiness, early cracking or occasional small lifting scales may be present); 3 (Generalised moderate powederiness and/or heavy cracking and lifting scales; 4 (Generalised heavy powederiness and/or heavy cracking and lifting scales); 5 (Generalised high cracking and lifting scales, eczematous change may be present, powederiness may be present but not prominent, may see bleeding crack); 6 (Generalised severe cracking, eczematous change may be present, bleeding cracks may be present, scale large may be beginning to disappear). Lower scores reflect less dry skin.
Time Frame: At Baseline and Day 5 (3 hours post last wash procedure)
Population: ITT population (N=48) was the primary population of analysis, which included all participants who were randomized and received at least one wash procedure, including sterile water, and had at least one post-baseline clinical assessment. Number of participants analyzed for this endpoint were part of the ITT population, evaluated on Day 5.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Test: Data of this arm included all allotted sides of the forearms of the participants where test product (0.09 ml of the cleanser) was applied during the study.
- Positive Control: Data of this arm included all allotted sides of the forearms of the participants where positive control (Soap bar) was applied during the study.
- Negative Control: Data of this arm included all allotted sides of the forearms of the participants where Negative control (0.09 ml of sterile water) was applied during the study.
- No Treatment: Data of this arm included all allotted sides of the forearms of the participants which were left untreated during the study.
Arm/Group | Test | Positive Control | Negative Control | No Treatment
Number analyzed (Participants) | 44 | 44 | 44 | 44
Score on a scale | 0.48 (0.284) | 0.91 (0.291) | 0.56 (0.290) | 0.63 (0.307)
Statistical Analysis 1: Comparison: Test vs Negative Control; The null hypothesis (non-inferiority setting) is that the population mean dryness for Test minus Baxter Sterile Water (negative control) is at least 0.25; Test type: Non-Inferiority — The non-Inferiority margin is set at 0.25. The upper limit of the 90% CI is less than this and hence NI is met; p = 0.1769, ANOVA — No adjustment for multiple comparisons was made; ANOVA model with change from baseline in examiner assessment on dryness as response and treatment, site as fixed effects; participant as random effect; Mean Difference (Net) = -0.077, 90% CI 2-sided [-0.1707 to 0.0169] — Difference is first named treatment minus second named treatment such that a negative difference favors first named treatment
Statistical Analysis 2: Comparison: Positive Control vs Negative Control; The null hypothesis is that the difference in population mean dryness is zero; Test type: Superiority — This is a superiority test setting; p < .0001, ANOVA — No adjustment for multiple comparisons was made; ANOVA model with change from baseline in examiner assessment on dryness as response and treatment, site as fixed effects;participant as random effect; Mean Difference (Net) = 0.350, 90% CI 2-sided [0.2565 to 0.4441] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Test vs Positive Control; The null hypothesis is that the difference in population mean dryness is zero; Test type: Superiority — This is a superiority test setting; p < .0001, ANOVA — No adjustment for multiple comparisons was made; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.427, 90% CI 2-sided [0.3333 to 0.5211] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Negative Control vs No Treatment; The null hypothesis is that the difference in population mean dryness is zero; Test type: Superiority — This is a superiority test setting; p = 0.2518, ANOVA — No adjustment for multiple comparisons was made; [statistical method as in outcome 1, analysis 2]; Mean Difference (Net) = 0.065, 90% CI 2-sided [-0.0287 to 0.1592] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Baseline in Visual Assessment of Redness at Day 5
Description: Skin redness was assessed by a trained examiner according to following the scoring scale: 0 (No redness); 1(Barely detectable redness); 2(Slight redness); 3 (Moderate redness); 4 (Heavy or substantial redness); 5 (Extreme redness); 6 (Severe Redness). Lower scores reflect less skin redness.
Time Frame: At Baseline and Day 5 (3 hours post last wash procedure)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Test: Data of this arm included all allotted sides of the forearms of the participants where test product (0.09 ml of the cleanser)was applied during the study.
- Negative Control: Data of this arm included all allotted sides of the forearms of the participants where Negative control (0.09 ml of sterile water ) was applied during the study.
Arm/Group | Test | Positive Control | Negative Control | No Treatment
Number analyzed (Participants) | 44 | 44 | 44 | 44
Score on a scale | 0.01 (0.075) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)

3. Secondary Outcome: Change From Baseline in Visual Assessment of Dryness at Day 2, 3, and 4
Description: as for outcome 1
Time Frame: At Baseline and Day 2, 3, and 4 (3 hours post last wash procedure)
Population: ITT population (N=48) was the primary population of analysis, which included all participants who were randomized and received at least one wash procedure, including sterile water, and had at least one post-baseline clinical assessment.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Reference (Unwashed Area): Data of this arm included all allotted sides of the forearms of the participants which were left untreated during the study.
Arm/Group | Test | Positive Control | Negative Control | Reference (Unwashed Area)
Number analyzed (Participants) | 48 | 48 | 48 | 48
Score on a scale
  Day 2 | 0.25 (0.253) | 0.46 (0.307) | 0.28 (0.251) | 0.31 (0.265)
  Day 3: number analyzed (Participants) | 45 | 45 | 45 | 45
  Day 3 | 0.37 (0.248) | 0.66 (0.298) | 0.38 (0.285) | 0.42 (0.260)
  Day 4: number analyzed (Participants) | 44 | 44 | 44 | 44
  Day 4 | 0.43 (0.255) | 0.76 (0.314) | 0.42 (0.240) | 0.55 (0.302)

4. Secondary Outcome: Change From Baseline in Visual Assessment of Redness at Day 2, 3, and 4
Description: as for outcome 2
Time Frame: At Baseline and Day 2, 3, and 4 (3 hours post last wash procedure)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Test | Positive Control | Negative Control | Reference (Unwashed Area)
Number analyzed (Participants) | 48 | 48 | 48 | 48
Score on a scale
  Day 2 | 0.06 (0.167) | 0.05 (0.154) | 0.01 (0.072) | 0.01 (0.072)
  Day 3: number analyzed (Participants) | 45 | 45 | 45 | 48
  Day 3 | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Day 4: number analyzed (Participants) | 44 | 44 | 44 | 48
  Day 4 | 0.00 (0.00) | 0.01 (0.075) | 0.00 (0.00) | 0.02 (0.151)

5. Secondary Outcome: Change From Baseline in Transepidermal Water Loss (TEWL) at Day 5
Description: TEWL was measured using Tewameter. TEWL measuring principle was based on water vapour gradient determination between two pairs of sensors placed at different distances perpendicularly to the skin. The probe was held in place on the skin for one measurement, for approximately 40 seconds (sec), to ensure that a stable value has been established. The first part of the measurement belonged to the equilibration phase. The values of the last 10 sec were averaged as the actual measurement values. An increase in TEWL values shows damage to the skin barrier function.
Time Frame: At Baseline and Day 5 (3 hours post last wash procedure)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/m^2/hr
Groups:
- Test Product: Data of this arm included all allotted sides of the forearms of the participants where test product (0.09 ml of the cleanser)was applied during the study..
Arm/Group | Test Product | Positive Control | Negative Control | No Treatment
Number analyzed (Participants) | 44 | 44 | 44 | 44
g/m^2/hr | 0.91 (2.118) | 1.95 (2.025) | 0.94 (1.714) | 0.53 (1.682)

6. Secondary Outcome: Change From Baseline in Skin Moisturisation at Day 5
Description: Corneometry was used to measure moisture content of stratum corneum using corneometer. The measuring principle was based on changes in the capacitance of the measuring head, functioning as a condensator. Between the gold conductors of the probe an electrical field was built which allowed the dielectricity of the stratum corneum to be measured. Because the dielectricity of the skin varies as a function of its water content, the stratum corneum moisturisation can be measured. The Corneometer probe was placed in contact with the skin of the paarticipant's test site for 1-2 seconds per measurement. The Corneometer measurements were taken and an average (mean) reading was calculated for each site and time point. Corneometer values lower than 30 instrumental units (i.u.) represents very dry skin, while values between 30 und 50 i.u are typically for dry skin on the forearm. An increase in Corneometer values, therefore, corresponds to a skin-moisturising effect.
Time Frame: At Baseline and Day 5 (3 hours post last wash procedure)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: i.u.
Arm/Group | Test | Positive Control | Negative Control | No Treatment
Number analyzed (Participants) | 44 | 44 | 44 | 44
i.u. | 2.35 (5.341) | -4.57 (5.368) | 2.13 (4.803) | 0.34 (3.729)

ADVERSE EVENTS:
Time Frame: Approximately 5 days
Description: All treatment emergent adverse events (AEs) were reported.
Groups:
- Overall Participants: Included all participants who applied any of the study products.
Arm/Group | Test | Positive Control | Negative Control | No Treatment | Overall Participants
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/48 | 0/48 | 0/48 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48 | 0/48 | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 4/48 | 4/48 | 4/48 | 2/48 | 6/48
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Test (N=48) | Positive Control (N=48) | Negative Control (N=48) | No Treatment (N=48) | Overall Participants (N=48)
FOOD POISONING (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 1
TOOTHACHE (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 1
APPLICATION SITE PRURITUS (General disorders) | 1 | 0 | 0 | 0 | 1
APPLICATION SITE PAIN (General disorders) | 0 | 1 | 2 | 0 | 2
THERMAL BURN (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-03-06): https://cdn.clinicaltrials.gov/large-docs/88/NCT03119688/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-26): https://cdn.clinicaltrials.gov/large-docs/88/NCT03119688/SAP_001.pdf